CLINICAL TRIAL: NCT03949608
Title: Randomized, Single Center Study About the Impact of an E-learning Dedicated to Myocardial Infarction Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Christel Bruggmann, PhD student and clinical pharmacist, University of Lausanne Hospitals
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-02223
Record Dates: First submitted 2019-04-25; First posted 2019-05-14 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Acute Myocardial Infarction
Keywords: e-learning; drug adherence; health literacy
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: We will randomize patients by block of 2 weeks of inclusion in intervention or controlled group. Each 2 weeks, all participants will be included in the intervention group, and the next 2 weeks the participants will be included in the control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BASIC (Experimental): "mon cœur, mon BASIC" video viewing and installation in the own smartphone or tablet of the patient
  Interventions: Other: E-learning
- Control (No Intervention): Usual care

INTERVENTIONS:
Other: E-learning — The intervention consists of the presentation and installation of an internet tool to educate the patient about his heart condition and about his medications in addition to usual care. The tool is an interactive web-hosting video called "Mon Coeur, mon BASIC" adaptable to smartphones and tablets. The total length of the video is around 15 minutes. The e-learning is interactive because of the possibility to click in the video to have more details about a particular point. The tool includes a part about the heart and particularly about the ACS (physiopathology, diagnosis, coronarography, angioplasty). A second part includes an education about the medications prescribed. The patient will select the medication being prescribed and receive information about it.
  Arms: BASIC

SUMMARY:
Acute coronary syndrome (ACS) is still one of the major cause of morbi-mortality in Europe. After an ACS, patients should be treated with secondary prevention medication to reduce the risk of recurrence. However, it is known that patients do not take all their medicines as expected, which leads to readmission at the hospital. To enhance drug adherence, the investigators sought to develop an interactive e-learning tool for these patients. This e-learning includes information about the disease, the acute care and the subsequent medications being prescribed. The tool is now ready to use and the investigators want to assess if it has the impact to enhance self-care management of ACS patients.

DETAILED DESCRIPTION:
Cardiovascular disease is a major cause of morbi-mortality in industrialized countries. Risk of recurrence after appropriate treatment is particularly frequent in patients with inadequate observance. Secondary prevention is therefore essential to reduce the morbi-mortality of high-risk cardiovascular patients. Risk factor control and lifestyle interventions are important for these high-risk patients to reduce the overall incidence of cardiac disease. To treat these risk factors and for secondary prevention after a cardiovascular event, some medications have been shown to be efficient and European guidelines have been written to enhance evidence-based medicine prescriptions for STEMI and NSTEMI. Despite this, concerns have been postulated about patient's self-adherence to these treatments. A study has shown a long-term adherence to medications of 71% for Aspirin, 46% for β-blockers and 44% for Lipid-lowering therapy for Coronary Artery Disease (CAD) patients. Non-adherence has been associated with increased morbi-mortality in this population.

Therefore, a variety of interventions was identified to enhance patient adherence to medication in the cardiovascular field. These strategies included:

* Informational intervention (mailed information)
* Sending reminder postcards, illustrated daily medication schedule distribution
* Counseling on the importance of adherence to their cardiovascular medication and review of each medication during the hospital stay
* Clinical pharmacist intervention with medication reconciliation, medication education, facilitation of the delivery of discharge medications, and post-discharge telephone call within 48-72h These interventions showed an impact on long-term medication adherence and health literacy, which could lead to an improvement of the morbi-mortality of cardiovascular risk patients.

In a previous study conducted at the University hospital of Lausanne, the investigators showed a very high prescription rate of guidelines-recommended medications for patients involved in the CHUV STEMI (ST-Elevation Myocardial Infarction) network. Therefore, the next step to reduce the morbi-mortality of high-risk cardiovascular patients is to enhance patient adherence to the cardiovascular drug regimen. Patient education is known as an effective process to enhance drug adherence. Unfortunately, patient education is difficult to implement because of it costs and for the time needed to educate the patient. The investigator's aim at testing a new approach using an e-learning tool for patient education purpose. The e-learning will be interactive and easy to use. It will inform the patient about his heart disease (acute coronary syndrome) and about his medications in a short time.

ELIGIBILITY:
Inclusion Criteria:

* Admission for acute coronary syndrome (ACS) in the cardiology unit of the University hospital of Lausanne (NSTEMI or STEMI)
* Have a percutaneous coronary intervention (PCI) as therapeutic strategy
* Patients going through an elective PCI for a second vessel after having suffered from an acute coronary syndrome in the previous month
* > 18 years
* Total discernment capacity and French speaking
* Have a digital tablet, a smartphone or a computer to have the possibility to watch the e-learning at home
* Informed Consent as documented by signature (Appendix Informed Consent Form)

Exclusion Criteria:

* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Refugee claimants, homeless persons, prisoners by impossibility to contact them after discharge
* Patients with communication problems
* Life expectancy < 6 months caused by other co-morbidities

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2020-03-22 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
ARMS (Adherence to Refill and Medication Score) score difference | 1,3 and 6 months
  Adherence to Refill and Medication Score is a self-reported questionnaire with 12-items. 8 items assess adherence to taking medications, and 4 items assess the refill to medication. The results can vary from 12 (most adherent) to 48 (less adherent). The ARMS questionnaire will be assessed after 1 month, 3 months and 6 months. We will assess the difference in the mean ARMS score between control group and intervention group at these 3 timepoints.

SECONDARY OUTCOMES:
Knowledge about the disease and medications | at time of inclusion, 1 day after inclusion for control group and after the viewing of the video for the intervention group, 1 month, 3 months and 6 months
  Difference in a knowledge score assessed with a 9 multiple choice questions about the disease (examples: what is a coronary artery? What happens during an acute myocardial infarction? Which medication is used to reduce cholesterol level?). The maximum score is 9 and the minimum is 0. The mean score will be tested between intervention and control group. The score variation will be assessed during time after ACS.
LDL-c measurement | 3 months
  Difference in LDL-c measurements from discharge to 3 months
BMI | 6 months
  Difference in BMI from discharge to 6 months
Target Blood Pressure | 6 months
  proportion of patients being in the target blood pressure measurements at 6 months
composite endpoint of readmission, reinfarction or emergency visit | 6 months
  Readmissions, reinfarction and emergency visit will be assessed with a questionnaire at 6 months. We will assess if there is a difference between intervention and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Christel Bruggmann, PharmD, Principal Investigator — Centre Hospitalier Universitaire Vaudois (CHUV)
Locations (1):
- Centre Hsopitalier Universitaire Vaudois, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bruggmann C, Adjedj J, Sardy S, Muller O, Voirol P, Sadeghipour F. Effects of the Interactive Web-Based Video "Mon Coeur, Mon BASIC" on Drug Adherence of Patients With Myocardial Infarction: Randomized Controlled Trial. J Med Internet Res. 2021 Aug 30;23(8):e21938. doi: 10.2196/21938. PMID 34459744